CLINICAL TRIAL: NCT01482715
Title: A Phase I/II, Open-Label, Safety, Pharmacokinetic, and Preliminary Efficacy Study of Oral Rucaparib in Patients With gBRCA Mutation Ovarian Cancer or Other Solid Tumor
Brief Title: A Study of Oral Rucaparib in Patients With a Solid Tumor (Phase I) or With gBRCA Mutation Ovarian Cancer (Phase II)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: pharmaand GmbH (Industry)
Collaborators: Foundation Medicine (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CO-338-010; 2011-004250-26 (EudraCT Number)
Record Dates: First submitted 2011-11-22; First posted 2011-11-30 (Estimated); Results first posted 2020-12-08 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Peritoneal Cancer; Advanced Solid Tumor With Evidence of Germline or Somatic BRCA
Keywords: gBRCA ovarian cancer; platinum sensitive; PARP Inhibitor; Rucaparib; CO-338; PF 01367338; AG 14699; BRCA1; BRCA2; platinum sensitive ovarian cancer; platinum sensitive gBRCA ovarian cancer; gynecological cancer; relapsed disease; homologous recombination deficiency; HRD
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Recurrence | interventions — rucaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Part 1 (Phase 1) (Experimental): Rucaparib 40, 80, 160, 300, 500 mg QD and 240, 360, 480, 600, 840 mg BID, for continuous 21-day cycles. Patients in Part 1 were initially treated in a Dose-escalation Evaluation Period (Cycle 1) and could then continue to receive treatment in an optional Treatment-extension Period (Cycle 2 and beyond).
  Interventions: Drug: Rucaparib
- Part 2A (Phase 2) (Experimental): Rucaparib 600 mg BID for 21-day cycles.
  Interventions: Drug: Rucaparib
- Part 2B (Phase 2) (Experimental): Rucaparib 600 mg BID for 21-day cycles.
  Interventions: Drug: Rucaparib
- Part 3 (Phase 2) (Experimental): Rucaparib 600 mg BID for 21-day cycles. Patients also received a single administration of 600 mg rucaparib on both Day -7 and Day 1 for assessing the effect of food on PK.
  Interventions: Drug: Rucaparib

INTERVENTIONS:
Drug: Rucaparib — Oral tablets administered daily with 8 oz (240 mL) of water on an empty stomach or with food; 21-day cycles of treatment. In Part 1, the initial dose level is 40 mg/day (once a day); doses and dosing frequency(e.g. twice a day or three times a day) will be adjusted until Maximum Tolerated Dose (MTD) and the Recommended Phase 2 Dose (RP2D) are established. Patients enrolled in Part 2 and Part 3 will receive the RP2D for continuous 21-day treatment cycles until disease progression.
  Other Names: CO-338; PF 01367338, AG 14699

SUMMARY:
Part 1 (Completed Enrollment) - The purpose of the first part of the study was to evaluate the safety of different doses and dosing regimens of oral rucaparib administered daily to patients with solid tumors.

Part 2A (Completed Enrollment) and Part 2B (Completed Enrollment) - The purpose of the second part of the study is to determine the safety and clinical activity of the RP2D of oral rucaparib administered daily to patients with a known deleterious BRCA mutation (germline or somatic).

Part 3 (Completed Enrollment) - The purpose of the third part of the study is to further evaluate PK of higher dose strength tablets at the RP2D in patients with any advanced solid tumor, inclusive of lymphoma, with evidence of a BRCA mutation (germline or somatic).

DETAILED DESCRIPTION:
Rucaparib (CO-338; formerly known as PF 01367338 and AG 14699) is an orally available, small molecule inhibitor of poly-adenosine diphosphate [ADP] ribose polymerase (PARP) being developed for treatment of ovarian cancer associated with homologous recombination [HR] DNA repair deficiency (HRD). The safety and efficacy of rucaparib has been evaluated in several Phase 1 and Phase 2 studies.

An oral formulation is the focus of current development efforts. Rucaparib is currently being investigated as monotherapy in patients with cancer associated with BRCA1 or BRCA2 mutations. For this study, it is anticipated that rucaparib will promote cell death in the BRCA-deficient tumor cells of ovarian cancer patients with evidence of a germline mutation, thereby limiting tumor progression and providing therapeutic benefit.

ELIGIBILITY:
The following eligibility criteria below pertain to patients enrolling into Part 2B of the study.

Inclusion Criteria:

* Have a known deleterious BRCA mutation (gBRCA or sBRCA) (as determined by a local laboratory that has received an international or country-specific, quality standards certification)
* Have evidence of measurable disease as defined by RECIST Version 1.1
* Have sufficient archival FFPE tumor tissue available for planned analyses. Archival tissue from the most recently collected biopsy or debulking surgery should be provided, if available.
* Have a histologically confirmed diagnosis of high-grade epithelial ovarian, fallopian tube, or primary peritoneal cancer
* Have received at least three prior chemotherapy regimens and have relapsed disease confirmed by radiologic assessment

Exclusion Criteria:

* Active second malignancy, i.e., patient known to have potentially fatal cancer present for which she may be (but not necessarily) currently receiving treatment

  a. Patients with a history of malignancy that has been completely treated, with no evidence of that cancer currently, are permitted to enroll in the trial provided all chemotherapy was completed >6 months prior and/or bone marrow transplant (BMT) >2 years prior to first dose of rucaparib
* Prior treatment with any PARP inhibitor.
* Untreated or symptomatic central nervous system (CNS) metastases. Patients with asymptomatic CNS metastases are eligible provided they have been clinically stable for at least 4 weeks.
* Received treatment with chemotherapy, radiation, antibody therapy or other immunotherapy, gene therapy, vaccine therapy, angiogenesis inhibitors, or experimental drugs 14 days prior to first dose of rucaparib and/or ongoing adverse effects from such treatment > NCI CTCAE Grade 1 (Grade 2 non-hematologic toxicity to most recent treatment may be permitted with prior advanced approval from Sponsor).
* Hospitalization for bowel obstruction within 3 months prior to enrollment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2011-11 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (16):
- United States (6):
  - UCSF, San Francisco, California
  - Sarah Cannon Research Institute, Sarasota, Florida
  - Dana-Farber Cancer Institute (Part 3 only), Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada
- Israel (2):
  - Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Hospital Vall d'Hebron, Barcelona, Spain
- United Kingdom (6):
  - Guy's and St Thomas NHS Foundation Trust, London, England
  - Royal Marsden NHS Foundation Trust, London, England
  - Imperial College Healthcare, London, England
  - Newcastle University, Newcastle upon Tyne, England
  - Institution of Cancer Science, University of Glasgow Wolfson Wohl Cancer Research, Glasgow, Scotland
  - University College London Cancer Institute, London

REFERENCES:
- [Derived] Kristeleit RS, Drew Y, Oza AM, Domchek SM, Banerjee S, Glasspool RM, Balmana J, Chen LM, Patel MR, Burris HA, Safra T, Borrow J, Lin KK, Goble S, Maloney L, Shapira-Frommer R. Efficacy and safety of rucaparib treatment in patients with BRCA-mutated, relapsed ovarian cancer: final results from Study 10. Br J Cancer. 2023 Jan;128(2):255-265. doi: 10.1038/s41416-022-02022-y. Epub 2022 Dec 8. PMID 36482193
- [Derived] Green ML, Ma SC, Goble S, Giordano H, Maloney L, Simmons AD, Beltman J, Harding TC, Xiao JJ. Population pharmacokinetics of rucaparib in patients with advanced ovarian cancer or other solid tumors. Cancer Chemother Pharmacol. 2022 May;89(5):671-682. doi: 10.1007/s00280-022-04413-7. Epub 2022 Apr 10. PMID 35397664
- [Derived] Kristeleit RS, Oaknin A, Ray-Coquard I, Leary A, Balmana J, Drew Y, Oza AM, Shapira-Frommer R, Domchek SM, Cameron T, Maloney L, Goble S, Lorusso D, Ledermann JA, McNeish IA. Antitumor activity of the poly(ADP-ribose) polymerase inhibitor rucaparib as monotherapy in patients with platinum-sensitive, relapsed, BRCA-mutated, high-grade ovarian cancer, and an update on safety. Int J Gynecol Cancer. 2019 Nov;29(9):1396-1404. doi: 10.1136/ijgc-2019-000623. PMID 31685558
- [Derived] Shapiro GI, Kristeleit RS, Burris HA, LoRusso P, Patel MR, Drew Y, Giordano H, Maloney L, Watkins S, Goble S, Jaw-Tsai S, Xiao JJ. Pharmacokinetic Study of Rucaparib in Patients With Advanced Solid Tumors. Clin Pharmacol Drug Dev. 2019 Jan;8(1):107-118. doi: 10.1002/cpdd.575. Epub 2018 May 25. PMID 29799676

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 15 investigative sites in the United States (6 sites), United Kingdom (5 sites), Spain (1 site), Israel (2 sites), and Canada (1 site).
Groups:
- Rucaparib 40 mg QD (Part 1): Rucaparib 40 mg once a day (QD) for continuous 21-day cycles
- Rucaparib 80 mg QD (Part 1): Rucaparib 80 mg once a day (QD) for continuous 21-day cycles
- Rucaparib 160 mg QD (Part 1): Rucaparib 160 mg once a day (QD) for continuous 21-day cycles
- Rucaparib 300 mg QD (Part 1): Rucaparib 300 mg once a day (QD) for continuous 21-day cycles
- Rucaparib 500 mg QD (Part 1): Rucaparib 500 mg once a day (QD) for continuous 21-day cycles
- Rucaparib 240 mg BID (Part 1): Rucaparib 240 mg twice a day (BID) for continuous 21-day cycles
- Rucaparib 360 mg BID (Part 1): Rucaparib 360 mg twice a day (BID) for continuous 21-day cycles
- Rucaparib 480 mg BID (Part 1): Rucaparib 480 mg twice a day (BID) for continuous 21-day cycles
- Rucaparib 600 mg BID (Part 1): Rucaparib 600 mg twice a day (BID) for continuous 21-day cycles
- Rucaparib 840 mg BID (Part 1): Rucaparib 840 mg twice a day (BID) for continuous 21-day cycles
- Rucaparib 600 mg BID (Part 2A); Rucaparib 600 mg BID (Part 2B): Rucaparib 600 mg twice a day (BID) for 21-day cycles
- Rucaparib 600 mg BID (Part 3): Rucaparib 600 mg twice a day (BID) for 21-day cycles. Patients also received a single administration of 600 mg rucaparib on both Day -7 and Day 1 for assessing the effect of food on PK.
Period: Overall Study
Arm/Group | Rucaparib 40 mg QD (Part 1) | Rucaparib 80 mg QD (Part 1) | Rucaparib 160 mg QD (Part 1) | Rucaparib 300 mg QD (Part 1) | Rucaparib 500 mg QD (Part 1) | Rucaparib 240 mg BID (Part 1) | Rucaparib 360 mg BID (Part 1) | Rucaparib 480 mg BID (Part 1) | Rucaparib 600 mg BID (Part 1) | Rucaparib 840 mg BID (Part 1) | Rucaparib 600 mg BID (Part 2A) | Rucaparib 600 mg BID (Part 2B) | Rucaparib 600 mg BID (Part 3)
Started | 6 | 3 | 4 | 9 | 4 | 3 | 8 | 9 | 7 | 3 | 42 | 12 | 26
Completed | 6 | 3 | 4 | 9 | 4 | 3 | 8 | 9 | 7 | 3 | 42 | 12 | 26
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Rucaparib 40 mg QD (Part 1): Rucaparib 40 mg QD for continuous 21-day cycles
- Rucaparib 80 mg QD (Part 1): Rucaparib 80 mg QD for continuous 21-day cycles
- Rucaparib 160 mg QD (Part 1): Rucaparib 160 mg QD for continuous 21-day cycles
- Rucaparib 300 mg QD (Part 1): Rucaparib 300 mg QD for continuous 21-day cycles
- Rucaparib 500 mg QD (Part 1): Rucaparib 500 mg QD for continuous 21-day cycles
- Rucaparib 240 mg BID (Part 1): Rucaparib 240 mg BID for continuous 21-day cycles
- Rucaparib 360 mg BID (Part 1): Rucaparib 360 mg BID for continuous 21-day cycles
- Rucaparib 480 mg BID (Part 1): Rucaparib 480 mg BID for continuous 21-day cycles
- Rucaparib 600 mg BID (Part 1); Rucaparib 600 mg BID (Part 2A); Rucaparib 600 mg BID (Part 2B); Rucaparib 600 mg BID (Part 3): Rucaparib 600 mg BID for continuous 21-day cycles
- Rucaparib 840 mg BID (Part 1): Rucaparib 840 mg BID for continuous 21-day cycles
- Total: Total of all reporting groups
Arm/Group | Rucaparib 40 mg QD (Part 1) | Rucaparib 80 mg QD (Part 1) | Rucaparib 160 mg QD (Part 1) | Rucaparib 300 mg QD (Part 1) | Rucaparib 500 mg QD (Part 1) | Rucaparib 240 mg BID (Part 1) | Rucaparib 360 mg BID (Part 1) | Rucaparib 480 mg BID (Part 1) | Rucaparib 600 mg BID (Part 1) | Rucaparib 840 mg BID (Part 1) | Rucaparib 600 mg BID (Part 2A) | Rucaparib 600 mg BID (Part 2B) | Rucaparib 600 mg BID (Part 3) | Total
Number analyzed (Participants) | 6 | 3 | 4 | 9 | 4 | 3 | 8 | 9 | 7 | 3 | 42 | 12 | 26 | 136
Age, Continuous [Median (Full Range); unit: years] | 63.5 [45.0 to 71.0] | 46.0 [41.0 to 49.0] | 52.0 [37.0 to 56.0] | 48.0 [41.0 to 63.0] | 29.5 [21.0 to 56.0] | 64.0 [62.0 to 68.0] | 49.5 [32.0 to 71.0] | 46.0 [28.0 to 70.0] | 52.0 [35.0 to 57.0] | 55.0 [42.0 to 59.0] | 56.5 [42.0 to 84.0] | 57.5 [46.0 to 72.0] | 59.5 [39.0 to 79.0] | 57.0 [21.0 to 84.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 4 | 9 | 2 | 2 | 7 | 9 | 7 | 2 | 42 | 12 | 21 | 126
  Male | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 5 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 3 | 0 | 1 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 2 | 9
  White | 6 | 3 | 4 | 7 | 3 | 3 | 6 | 8 | 7 | 2 | 35 | 11 | 22 | 117
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate Per RECIST Version 1.1 (Part 2)
Description: The confirmed response rate by RECIST v1.1 is defined as the proportion of patients with a confirmed Complete Response (CR) or Partial Response (PR) on subsequent tumor assessment at least 28 days after first response documentation.
Time Frame: Time from first dose to date of progression, up to approximately 8 months
Population: Efficacy-Evaluable Population - all Part 2 patients who met eligibility criteria, received at least 1 dose of rucaparib, had measurable tumor lesions at baseline, and had at least 1 post-baseline disease assessment. 2 patients in Part 2A discontinued treatment due to an AE and did not have a post-baseline disease assessment.
Measure: Count of Participants; unit: Participants
Groups:
- Rucaparib 600 mg BID (Part 2A); Rucaparib 600 mg BID (Part 2B): Rucaparib 600 mg BID for 21-day cycles
Arm/Group | Rucaparib 600 mg BID (Part 2A) | Rucaparib 600 mg BID (Part 2B)
Number analyzed (Participants) | 40 | 12
Participants | 25 | 7

2. Primary Outcome: Number of Participants With a Dose Limiting Toxicity (DLT)
Description: The number of Part 1 (Phase 1) patients who experienced dose limiting toxicities after one cycle (21 days) of study drug.
Time Frame: Cycle 1 Day 1 to Cycle 1 Day 21
Population: DLT-evaluable population - all patients enrolled into Part 1 of the study who received at least 17 complete days of rucaparib and completed Cycle 1 of treatment, or who experienced a DLT in Cycle 1.
Measure: Count of Participants; unit: Participants
Groups:
- Rucaparib 40 mg QD (Part 1): Rucaparib 40 mg once a day (QD)
- Rucaparib 80 mg QD (Part 1): Rucaparib 80 mg once a day (QD)
- Rucaparib 160 mg QD (Part 1): Rucaparib 160 mg once a day (QD)
- Rucaparib 300 mg QD (Part 1): Rucaparib 300 mg once a day (QD)
- Rucaparib 500 mg QD (Part 1): Rucaparib 500 mg once a day (QD)
- Rucaparib 240 mg BID (Part 1): Rucaparib 240 mg twice a day (BID)
- Rucaparib 360 mg BID (Part 1): Rucaparib 360 mg twice a day (BID)
- Rucaparib 480 mg BID (Part 1): Rucaparib 480 mg twice a day (BID)
- Rucaparib 600 mg BID (Part 1): Rucaparib 600 mg twice a day (BID)
- Rucaparib 840 mg BID (Part 1): Rucaparib 840 mg twice a day (BID)
Arm/Group | Rucaparib 40 mg QD (Part 1) | Rucaparib 80 mg QD (Part 1) | Rucaparib 160 mg QD (Part 1) | Rucaparib 300 mg QD (Part 1) | Rucaparib 500 mg QD (Part 1) | Rucaparib 240 mg BID (Part 1) | Rucaparib 360 mg BID (Part 1) | Rucaparib 480 mg BID (Part 1) | Rucaparib 600 mg BID (Part 1) | Rucaparib 840 mg BID (Part 1)
Number analyzed (Participants) | 6 | 3 | 4 | 9 | 4 | 3 | 8 | 9 | 7 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Rucaparib 40 mg QD (Part 1) vs Rucaparib 80 mg QD (Part 1) vs Rucaparib 160 mg QD (Part 1) vs Rucaparib 300 mg QD (Part 1) vs Rucaparib 500 mg QD (Part 1) vs Rucaparib 240 mg BID (Part 1) vs Rucaparib 360 mg BID (Part 1) vs Rucaparib 480 mg BID (Part 1) vs Rucaparib 600 mg BID (Part 1) vs Rucaparib 840 mg BID (Part 1); Test type: Other; RP2D = 600; A MTD was not established based on observation of DLTs in Cycle 1 of treatment. The 600 mg BID dose was considered to be the maximum dose with an acceptable toxicity profile that could be continuously administered to patients and was selected as the recommended Phase 2 dose (RP2D)

3. Primary Outcome: PK Profile of Rucaparib - Cmax (Part 1)
Description: Cmax = maximum concentration following administration of rucaparib
Time Frame: Cycle 1 Day 1 to Cycle 1 Day 15, or approximately 15 days
Population: PK-evaluable population - all patients enrolled into Part 1 of the study who received at least one dose of rucaparib and had adequate PK assessments drawn for determination of the PK profile. For some arms, the number analyzed at Day 1 and Day 15 differs from the overall number based on number of evaluable samples collected at each time point.
Measure: Median (Full Range); unit: ng/mL
Groups:
- Rucaparib 40 mg QD: Rucaparib 40 mg once a day (QD)
- Rucaparib 80 mg QD: Rucaparib 80 mg once a day (QD)
- Rucaparib 160 mg QD: Rucaparib 160 mg once a day (QD)
- Rucaparib 300 mg QD: Rucaparib 300 mg once a day (QD)
- Rucaparib 500 mg QD: Rucaparib 500 mg once a day (QD)
- Rucaparib 240 mg BID: Rucaparib 240 mg twice a day (BID)
- Rucaparib 360 mg BID: Rucaparib 360 mg twice a day (BID)
- Rucaparib 480 mg BID: Rucaparib 480 mg twice a day (BID)
- Rucaparib 600 mg BID: Rucaparib 600 mg twice a day (BID)
- Rucaparib 840 mg BID: Rucaparib 840 mg twice a day (BID)
Arm/Group | Rucaparib 40 mg QD | Rucaparib 80 mg QD | Rucaparib 160 mg QD | Rucaparib 300 mg QD | Rucaparib 500 mg QD | Rucaparib 240 mg BID | Rucaparib 360 mg BID | Rucaparib 480 mg BID | Rucaparib 600 mg BID | Rucaparib 840 mg BID
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 3 | 3 | 8 | 9 | 7 | 3
ng/mL
  Day 1 Cmax | 120 [98.9 to 168] | 119 [65.7 to 158] | 255 [107 to 426] | 700 [368 to 818] | 699 [629 to 1520] | 132 [123 to 401] | 603 [244 to 1170] | 1090 [312 to 2440] | 972 [271 to 1790] | 954 [705 to 2470]
  Day 15 Cmax: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 8 | 7 | 2
  Day 15 Cmax | 159 [80.7 to 174] | 180 [108 to 237] | 267 [217 to 380] | 439 [340 to 1300] | 1250 [1170 to 1750] | 783 [619 to 1510] | 1220 [728 to 2320] | 2480 [922 to 6870] | 2330 [477 to 3670] | 3030 [3000 to 3060]

4. Primary Outcome: PK Profile of Rucaparib - Tmax (Part 1)
Description: Tmax = time to maximum concentration following administration of rucaparib
Time Frame: Cycle 1 Day 1 to Cycle 1 Day 15, or approximately 15 days
Population: as for outcome 3
Measure: Median (Full Range); unit: hr
Arm/Group | Rucaparib 40 mg QD | Rucaparib 80 mg QD | Rucaparib 160 mg QD | Rucaparib 300 mg QD | Rucaparib 500 mg QD | Rucaparib 240 mg BID | Rucaparib 360 mg BID | Rucaparib 480 mg BID | Rucaparib 600 mg BID | Rucaparib 840 mg BID
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 3 | 3 | 8 | 9 | 7 | 3
hr
  Day 1 Tmax | 2.5 [1 to 4] | 1.5 [1 to 2.5] | 4 [4 to 6.05] | 2.5 [1 to 4.08] | 4 [4 to 4] | 6 [4.05 to 6] | 3.23 [1.5 to 6] | 2.5 [1.5 to 4] | 4 [2.42 to 10] | 4 [2.5 to 8]
  Day 15 Tmax: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 8 | 7 | 2
  Day 15 Tmax | 4 [1 to 4.05] | 2.5 [2.5 to 2.57] | 3.75 [2.5 to 4] | 2.53 [2.5 to 8] | 4 [4 to 4.17] | 1.5 [1 to 4] | 3.3 [0 to 6.33] | 1.51 [0 to 6] | 4 [2.53 to 10] | 4.04 [4 to 4.07]

5. Primary Outcome: PK Profile of Rucaparib - AUC Last (Part 1)
Description: AUC last = Area under the plasma concentration-time curve from time 0 to the last recorded observation
Time Frame: Cycle 1 Day 1 to Cycle 1 Day 15, or approximately 15 days
Population: as for outcome 3
Measure: Median (Full Range); unit: hr*ng/mL
Arm/Group | Rucaparib 40 mg QD | Rucaparib 80 mg QD | Rucaparib 160 mg QD | Rucaparib 300 mg QD | Rucaparib 500 mg QD | Rucaparib 240 mg BID | Rucaparib 360 mg BID | Rucaparib 480 mg BID | Rucaparib 600 mg BID | Rucaparib 840 mg BID
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 3 | 3 | 8 | 9 | 7 | 3
hr*ng/mL
  Day 1 AUC last: number analyzed (Participants) | 2 | 3 | 4 | 3 | 3 | 3 | 8 | 9 | 7 | 3
  Day 1 AUC last | 915 [850 to 981] | 916 [555 to 930] | 2730 [1520 to 5230] | 5820 [3540 to 7860] | 7670 [6640 to 18700] | 875 [835 to 2430] | 4160 [1060 to 6670] | 6190 [1270 to 17200] | 6700 [1650 to 10900] | 5930 [5140 to 16700]
  Day 15 AUC last: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 8 | 7 | 2
  Day 15 AUC last | 2270 [889 to 2280] | 1870 [1340 to 2000] | 3510 [3130 to 5670] | 6090 [4020 to 18700] | 16500 [13900 to 29200] | 6340 [5100 to 12600] | 9110 [5950 to 17200] | 19400 [7480 to 55100] | 19700 [3090 to 32600] | 24900 [24100 to 25700]

6. Secondary Outcome: Progression-free Survival (PFS) According to RECIST v1.1, as Assessed by the Investigator (Part 2)
Description: PFS is calculated as 1+ the number of days from the first dose of study drug to disease progression by RECIST, as determined by the investigator or death due to any cause, whichever occurs first.
Time Frame: Cycle 1 Day 1 to End of Treatment, up to approximately 51 months
Population: Safety population: Consist of all Part 2 patients who received at least one dose of rucaparib
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Rucaparib 600 mg BID (Part 2A) | Rucaparib 600 mg BID (Part 2B)
Number analyzed (Participants) | 42 | 12
Days | 260 [203 to 373] | 280 [40 to 551]

7. Secondary Outcome: Duration of Response Per RECIST Version 1.1 (Part 2)
Description: Duration of response (DOR) for any confirmed RECIST CR or PR measured from the date of the first occurrence of a response until the first occurrence of PD per RECIST. For patients who continued treatment post-progression, the first date of progression was used for the analysis. Any patients with an ongoing response were censored at the date of the last post-baseline scan.
Time Frame: Cycle 1 Day 1 to End of Treatment, up to approximately 48 months
Population: Safety population - all Part 2 patients with confirmed response per investigator.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Rucaparib 600 mg BID (Part 2A) | Rucaparib 600 mg BID (Part 2B)
Number analyzed (Participants) | 25 | 7
Days | 270 [170 to 393] | 318 [106 to 497]

8. Secondary Outcome: Overall Survival (Part 2B)
Description: Overall survival (OS) is defined as the number of days from the date of first dose of study drug to the date of death, due to any cause. Patients without a documented event of death will be censored on the date of their last visit.
Time Frame: Cycle 1 Day 1 to date of death, assessed up to 38 months
Population: Safety population: Consist of all Part 2B patients who received at least one dose of rucaparib
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Rucaparib 600 mg BID (Part 2B)
Number analyzed (Participants) | 12
Days | 764 [166 to NA] — The upper confidence of the median is not reached due to not enough death events.

9. Secondary Outcome: Food Effect on PK of Rucaparib - Cmax (Part 1 and Part 3)
Description: Cmax = maximum concentration following administration of rucaparib. The effect of food on rucaparib PK parameters was assessed over a 24-hour period in blood samples from a subset of patients. Patients were given a single dose of 40 mg or 300 mg rucaparib (Part 1), or 600 mg rucaparib (Part 3) and were randomized to one of two sequences where they were either Fed (with a high-fat meal) or Fasted (without a high-fat meal) on Day -7 or Cycle 1 Day 1. On each day, patients underwent blood sampling for PK at the specified time points. The median Fed and Fasted Cmax values were calculated for each arm.
Time Frame: Day -7 to Cycle 1 Day 1, or approximately 7 days
Population: A subset of patients treated with either 40 mg, 300 mg, or 600 mg rucaparib
Measure: Median (Full Range); unit: ng/mL
Groups:
- Rucaparib 40 mg QD: Rucaparib 40 mg single dose
- Rucaparib 300 mg QD: Rucaparib 300 mg single dose
- Rucaparib 600 mg BID: Rucaparib 600 mg single dose
Arm/Group | Rucaparib 40 mg QD | Rucaparib 300 mg QD | Rucaparib 600 mg BID
Number analyzed (Participants) | 3 | 6 | 26
ng/mL
  Cmax Fasted | 57.6 [45.2 to 131] | 424 [182 to 638] | 585 [127 to 3100]
  Cmax Fed | 71.1 [21.3 to 102] | 393 [177 to 1210] | 746 [198 to 2640]

10. Secondary Outcome: Food Effect on PK of Rucaparib - Tmax (Part 1 and Part 3)
Description: Tmax = time to maximum concentration following administration of rucaparib. The effect of food on rucaparib PK parameters was assessed over a 24-hour period in blood samples from a subset of patients. Patients were given a single dose of 40 mg or 300 mg rucaparib (Part 1), or 600 mg rucaparib (Part 3) and were randomized to one of two sequences where they were either Fed (with a high-fat meal) or Fasted (without a high-fat meal) on Day -7 or Cycle 1 Day 1. On each day, patients underwent blood sampling for PK at the specified time points. The median Fed and Fasted Tmax values were calculated for each arm.
Time Frame: Day -7 to Cycle 1 Day 1, or approximately 7 days
Population: A subset of patients treated with either 40 mg, 300 mg, or 600 mg rucaparib
Measure: Median (Full Range); unit: hr
Arm/Group | Rucaparib 40 mg QD | Rucaparib 300 mg QD | Rucaparib 600 mg BID
Number analyzed (Participants) | 3 | 6 | 26
hr
  Tmax Fasted | 4 [2.5 to 4.05] | 4.09 [2.5 to 24.22] | 4.02 [0.53 to 24.83]
  Tmax Fed | 2.55 [1 to 4.08] | 5.95 [2.53 to 10] | 7.83 [1.5 to 24.45]

11. Secondary Outcome: Food Effect on PK of Rucaparib - AUC Last (Part 1 and Part 3)
Description: AUC last = Area under the plasma concentration-time curve from time 0 to the last recorded observation. The effect of food on rucaparib PK parameters was assessed over a 24-hour period in blood samples from a subset of patients. Patients were given a single dose of 40 mg or 300 mg rucaparib (Part 1), or 600 mg rucaparib (Part 3) and were randomized to one of two sequences where they were either Fed (with a high-fat meal) or Fasted (without a high-fat meal) on Day -7 or Cycle 1 Day 1. On each day, patients underwent blood sampling for PK at the specified time points. The median Fed and Fasted AUC last values were calculated for each arm.
Time Frame: Day -7 to Cycle 1 Day 1, or approximately 7 days
Population: A subset of patients treated with either 40 mg, 300 mg, or 600 mg rucaparib. For the 40 mg and 300 mg arms, the number analyzed at Day 1 and Day 15 differs from the overall number based on number of evaluable samples collected at each time point.
Measure: Median (Full Range); unit: hr*ng/mL
Arm/Group | Rucaparib 40 mg QD | Rucaparib 300 mg QD | Rucaparib 600 mg BID
Number analyzed (Participants) | 3 | 6 | 26
hr*ng/mL
  AUC last Fasted | 468 [347 to 1410] | 5410 [2390 to 8680] | 7050 [1110 to 33000]
  AUC last Fed: number analyzed (Participants) | 2 | 5 | 26
  AUC last Fed | 794 [415 to 1170] | 6000 [2670 to 12100] | 10900 [1990 to 40400]

12. Secondary Outcome: QTcF Value Change From Baseline (Part 1)
Description: QTcF value change from baseline by daily dose corrected using Fridericia's method (QTcF). To evaluate the effects of rucaparib on the QT (interval from Q wave to T wave)/QTc (interval corrected for heart rate) interval, all patients underwent serial ECG monitoring at Screening, on Cycle 1 Day -1, Cycle 1 Day 1, Cycle 1 Day 15, Cycle 1 Day 22, on Day 1 of all subsequent cycles, at the EOT Visit, and as clinically indicated. Worst post-baseline QTcF value was used to categorize each patient.
Time Frame: Screening to End of Treatment, up to approximately 15 months
Population: Safety population: Consist of all Part 1 patients who received at least one dose of rucaparib. One patient in the 40 mg dose group had no Baseline evaluation and was excluded from analyses of change from Baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Rucaparib 40 mg QD | Rucaparib 80 mg QD | Rucaparib 160 mg QD | Rucaparib 300 mg QD | Rucaparib 500 mg QD | Rucaparib 240 mg BID | Rucaparib 360 mg BID | Rucaparib 480 mg BID | Rucaparib 600 mg BID | Rucaparib 840 mg BID
Number analyzed (Participants) | 5 | 3 | 4 | 9 | 4 | 3 | 8 | 9 | 7 | 3
Participants
  QTcF Change from Baseline <30 msec | 5 | 3 | 4 | 9 | 3 | 3 | 8 | 9 | 7 | 3
  QTcF Change from Baseline ≥30 to <60 msec | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  QTcF Change from Baseline ≥60 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were reported from the date of first dose of study drug and within 28 days after last dose of study drug. The first patient was dosed in 2012 through study completion in 2017, with an average treatment duration of 173.9 days in Part 1, 331.1 days in Part 2A, 348.2 days in Part 2B, and 198.8 days in Part 3.
Groups:
- Rucaparib 40 mg QD (Part 1): Rucaparib 40 mg QD for 21-day cycles
- Rucaparib 80 mg QD (Part 1): Rucaparib 80 mg QD for 21-day cycles
- Rucaparib 160 mg QD (Part 1): Rucaparib 160 mg QD for 21-day cycles
- Rucaparib 300 mg QD (Part 1): Rucaparib 300 mg QD for 21-day cycles
- Rucaparib 500 mg QD (Part 1): Rucaparib 500 mg QD for 21-day cycles
- Rucaparib 240 mg BID (Part 1): Rucaparib 240 mg BID for 21-day cycles
- Rucaparib 360 mg BID (Part 1): Rucaparib 360 mg BID for 21-day cycles
- Rucaparib 480 mg BID (Part 1): Rucaparib 480 mg BID for 21-day cycles
- Rucaparib 600 mg BID (Part 1); Rucaparib 600 mg BID (Part 2A); Rucaparib 600 mg BID (Part 2B); Rucaparib 600 mg BID (Part 3): Rucaparib 600 mg BID for 21-day cycles
- Rucaparib 840 mg BID (Part 1): Rucaparib 840 mg BID for 21-day cycles
Arm/Group | Rucaparib 40 mg QD (Part 1) | Rucaparib 80 mg QD (Part 1) | Rucaparib 160 mg QD (Part 1) | Rucaparib 300 mg QD (Part 1) | Rucaparib 500 mg QD (Part 1) | Rucaparib 240 mg BID (Part 1) | Rucaparib 360 mg BID (Part 1) | Rucaparib 480 mg BID (Part 1) | Rucaparib 600 mg BID (Part 1) | Rucaparib 840 mg BID (Part 1) | Rucaparib 600 mg BID (Part 2A) | Rucaparib 600 mg BID (Part 2B) | Rucaparib 600 mg BID (Part 3)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/3 | 1/4 | 1/9 | 0/4 | 1/3 | 0/8 | 1/9 | 0/7 | 0/3 | 4/42 | 1/12 | 4/26
Serious Adverse Events (participants affected / at risk) | 2/6 | 1/3 | 3/4 | 4/9 | 0/4 | 2/3 | 3/8 | 4/9 | 1/7 | 1/3 | 19/42 | 3/12 | 9/26
Other Adverse Events (participants affected / at risk) | 6/6 | 3/3 | 4/4 | 9/9 | 4/4 | 3/3 | 8/8 | 8/9 | 7/7 | 3/3 | 41/42 | 12/12 | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rucaparib 40 mg QD (Part 1) (N=6) | Rucaparib 80 mg QD (Part 1) (N=3) | Rucaparib 160 mg QD (Part 1) (N=4) | Rucaparib 300 mg QD (Part 1) (N=9) | Rucaparib 500 mg QD (Part 1) (N=4) | Rucaparib 240 mg BID (Part 1) (N=3) | Rucaparib 360 mg BID (Part 1) (N=8) | Rucaparib 480 mg BID (Part 1) (N=9) | Rucaparib 600 mg BID (Part 1) (N=7) | Rucaparib 840 mg BID (Part 1) (N=3) | Rucaparib 600 mg BID (Part 2A) (N=42) | Rucaparib 600 mg BID (Part 2B) (N=12) | Rucaparib 600 mg BID (Part 3) (N=26)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Obstruction gastric (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cytomegalovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Epiglottiis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Urinary tract stoma complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
B-cell type acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 2 | 0 | 2 | 1 | 1 | 0 | 0 | 4 | 1 | 3
Myodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Vaginal fistula (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rucaparib 40 mg QD (Part 1) (N=6) | Rucaparib 80 mg QD (Part 1) (N=3) | Rucaparib 160 mg QD (Part 1) (N=4) | Rucaparib 300 mg QD (Part 1) (N=9) | Rucaparib 500 mg QD (Part 1) (N=4) | Rucaparib 240 mg BID (Part 1) (N=3) | Rucaparib 360 mg BID (Part 1) (N=8) | Rucaparib 480 mg BID (Part 1) (N=9) | Rucaparib 600 mg BID (Part 1) (N=7) | Rucaparib 840 mg BID (Part 1) (N=3) | Rucaparib 600 mg BID (Part 2A) (N=42) | Rucaparib 600 mg BID (Part 2B) (N=12) | Rucaparib 600 mg BID (Part 3) (N=26)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 3 | 1 | 0 | 4 | 3 | 4 | 1 | 30 | 8 | 6
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 2 | 0 | 9 | 2 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 8 | 4 | 3
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0
Conjunctival hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 3 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 2 | 2 | 1 | 0 | 11 | 0 | 4
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 5 | 0 | 0 | 2 | 3 | 1 | 1 | 20 | 5 | 4
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 1 | 1 | 5 | 2 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 2 | 5 | 0 | 0 | 3 | 2 | 1 | 0 | 22 | 7 | 7
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 0 | 2 | 0 | 1 | 1 | 2 | 2 | 3 | 17 | 3 | 4
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 3 | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 1 | 0 | 0 | 3 | 2 | 6
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 5 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 2 | 2
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 1 | 3 | 6 | 0 | 0 | 6 | 4 | 4 | 3 | 35 | 11 | 11
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 7 | 1 | 0
Tooth disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 3 | 4 | 1 | 0 | 3 | 5 | 4 | 2 | 24 | 9 | 9
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 13 | 1 | 2
Axillary pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 1 | 0
Early satiety (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 1 | 6 | 2 | 1 | 6 | 5 | 5 | 1 | 30 | 6 | 14
Influenza like illness (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 1 | 0
Injection site bruising (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 2
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 5
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 2
Pyrexia (General disorders) | 0 | 0 | 0 | 3 | 0 | 1 | 3 | 1 | 0 | 0 | 5 | 3 | 3
Allergy to arthropod bite (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 4 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 12 | 2 | 2
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 3 | 0 | 8 | 3 | 5
Viral upper respiratory infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 5 | 1 | 24 | 2 | 6
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 3 | 5 | 1 | 22 | 2 | 6
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 4 | 0 | 10 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 1 | 0
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 1 | 0 | 3 | 2 | 3
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 15 | 6 | 3
Blood potassium increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Blood urea increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 3 | 1 | 0 | 3 | 0 | 3
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 7 | 2 | 2
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 2
Weight decreased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 8 | 1 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 0 | 5 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 3 | 0 | 0 | 6 | 0 | 2 | 3 | 1 | 0 | 1 | 12 | 3 | 10
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 3 | 1 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 4 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 2 | 0 | 1 | 1 | 1 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 4 | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 7 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 5 | 2 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 3 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 9 | 3 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 0 | 7 | 2 | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 2 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 2 | 1 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 3 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 5 | 1 | 2
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 2 | 2 | 2 | 0 | 9 | 1 | 6
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 1 | 2 | 17 | 2 | 5
Headache (Nervous system disorders) | 2 | 0 | 1 | 2 | 0 | 0 | 2 | 0 | 2 | 1 | 20 | 2 | 2
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 1
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 6 | 0 | 2
Depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 4 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 1 | 1 | 0 | 6 | 0 | 2
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 3 | 0 | 2
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 3 | 2 | 2 | 10 | 2 | 4
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 3 | 3 | 1 | 1 | 11 | 1 | 4
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 3 | 0 | 0
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 1 | 1 | 0 | 7 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 8 | 1 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 6 | 1 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 2 | 1 | 0 | 5 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 6 | 1 | 3
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 8 | 1 | 3
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hot flush (Vascular disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 4 | 2 | 1
Lymphoedema (Vascular disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 5 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Splenomegaly (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Ear congestion (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Macular degeneration (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mydriasis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anal pruritus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Tongue ulceration (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth erosion (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Catheter site inflammation (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Local swelling (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nodule (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0
Suprapubic pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Ulcer (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hepatomegaly (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Furuncle (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Herpes virus infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Oral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Skin candida (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection enterococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood magnesium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood phosphorus decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood urea nitrogen/creatinine ratio increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Breath sounds abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Heart rate increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0
Bone lesion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Extremity contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sensory loss (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mental fatigue (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Obstructive uropathy (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pruritus genital (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vaginal fistula (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal discomfort (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catarrh (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypertrichosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor's agreements with investigators require proposed public disclosures of trial results to be submitted to Sponsor for review prior to publication. Sponsor may request deletion of confidential information or a delay in publication to address intellectual property concerns, but Sponsor may not suppress publication of the trial results indefinitely. Sponsor may request delay of a single-center publication until after the release of a multi-site publication or an agreed upon period of time.

DOCUMENTS (2):
  • Study Protocol (2016-06-29): https://cdn.clinicaltrials.gov/large-docs/15/NCT01482715/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-10): https://cdn.clinicaltrials.gov/large-docs/15/NCT01482715/SAP_001.pdf